CLINICAL TRIAL: NCT00934518
Title: Image Guided Intensity Modulated Reirradiation With Concurrent Cetuximab in the Treatment of Locoregionally Confined Relapsed Squamous Cell Carcinoma of the Head and Neck
Brief Title: Image Guided Intensity Modulated Reirradiation (IG-IMRT) With Cetuximab for Locoregionally Confined Recurrent Head and Neck Squamous Cell Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate patient accrual
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Heath Mackley, Associate Professor, Penn State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSHCI 08-066
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Squamous Cell Cancer of the Head and Neck
Keywords: Squamous cell carcinoma, Head and Neck cancer
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms | interventions — Radiation; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation and Cetuximab (Experimental): Radiation Therapy 60 Gy total dose in 30 fractions: 2.0 Gy/fraction once daily five fractions per week
  Cetuximab 400 mg/m2 of body surface area over a period of 120 minutes day 1 250 mg/m2 of body surface area over a period of 60 minutes weekly during radiation
  Interventions: Radiation: Radiation; Drug: Cetuximab

INTERVENTIONS:
Radiation: Radiation — Radiation Therapy 60 Gy total dose in 30 fractions: 2.0 Gy/fraction once daily five fractions per week
Drug: Cetuximab — Radiation Therapy 60 Gy total dose in 30 fractions: 2.0 Gy/fraction once daily five fractions per week
  Cetuximab 400 mg/m2 of body surface area over a period of 120 minutes day 1 250 mg/m2 of body surface area over a period of 60 minutes weekly during radiation

SUMMARY:
The standard treatment for head and neck cancer relapses in previously irradiated patients is controversial. Reirradiation has had some success, but many patients still die from their disease. Cetuximab is helpful in relapsed head and neck cancer, and it improves the effectiveness of radiation in some head and neck cancer patients. But, it has not been studied with reirradiation. The purpose of this study is to see the effects, both good and bad, of reirradiation with cetuximab.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a pathologically confirmed recurrence (reappearance of previously cleared) squamous cell cancer in the upper aerodigestive tract or a second squamous cell primary. Patients may have experienced more than one recurrence as long as the first recurrence occurred ≥6 months following the end of the prior RT.
* The recurrence or second primary must be confined to the head and neck above the clavicles (loco-regional recurrence).
* The majority (≥75%) of the tumor volume must have been in areas previously irradiated to ≥45 Gy. The previous irradiation must not exceed a maximum of 75 Gy.
* Patients must be at least 6 months from prior radiation therapy.
* If a resection is performed after the diagnosis of recurrence and before enrollment, either microscopic or macroscopic disease must be present (i.e. positive margins or gross residual).
* Karnofsky Performance Status 60-100.
* Granulocytes ≥ 1500/mm3, platelets ≥ 100,000/mm3, bilirubin ≤ 1.5 mg/dl, creatinine ≤ 1.5 mg/dl, within 6 weeks prior to registration.
* Must be able to submit previous radiation records (simulation and portal film if available) in order to assure that cord tolerance is not exceeded.
* Patients must sign a study-specific informed consent form prior to study entry.
* The patient must be between the ages of 18 and 75.

Exclusion Criteria:

* Distant metastases.
* Completely resected recurrence with negative margins.
* Other concurrent invasive malignancies.
* Prior invasive malignancy unless disease free for at least two years (prior in situ malignancies are permissible).
* Intercurrent medical illnesses which would impair patient tolerance to therapy or limit survival.
* Pregnant and nursing women are excluded because of the potential teratogenic effects and potential unknown effects on nursing newborns.
* Previous treatment with cetuximab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To estimate the incidence rate of acute and late toxicities associated with combined cetuximab and image guided intensity modulated reirradiation in patients with recurrent squamous cell cancer of the head and neck. | 5 years

SECONDARY OUTCOMES:
To estimate the median and one-year, disease-free, and overall survival rates of the treated patients. | 5 years
To determine the pattern of disease progression in treated patients. | 5 years
To identify the impact of cetuximab and image guided intensity modulated reirradiation on patients' quality of life. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Heath B Mackley, MD, Principal Investigator — Penn State Hershey Cancer Institute
Locations (1):
- Penn State Hershey Cancer Institute, Hershey, Pennsylvania, United States